CLINICAL TRIAL: NCT03784924
Title: EDRN Prostate MRI Biomarker Study and Reference Set
Brief Title: EDRN Prostate MRI Biomarker Study
Acronym: P-MRI
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); University of Alabama at Birmingham (Other); University of Chicago (Other); Cornell University (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Vanderbilt University (Other); Emory University (Other); University of Miami (Other); University of Texas (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, John Wei, David A Bloom Professor of Urology, Medical Director of Brighton Center for Specialty Care and Professor of Urology, Medical School, University of Michigan
Other Study IDs: 430
Record Dates: First submitted 2018-12-04; First posted 2018-12-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: PSA; Prostate Cancer
Keywords: Prostate cancer; psa; early detection; MRI
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 8 x 250ul and 10 x 100ul Serum 10 x 200ul EDTA Plasma
  1 x 500ul Buffy Coat
  1 x 1ml Whole Blood from EDTA Tube 2 x 5.0ml Unprocessed Raw Urine 4 x 5.0ml Whole Urine 4 x 5ml Supernatant
  1 x 50ul Pellet/Sediment FFPE tumor tissue (blocks) from all cancer foci Nitrocellulose tissue prints from all cores
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Initial prostate biopsy: Men who have never had a prostate biopsy, but have an elevated risk for prostate cancer such as elevated PSA who are scheduled or considered candidate for an initial prostate biopsy.
  Interventions: Diagnostic Test: MRI prostate

INTERVENTIONS:
Diagnostic Test: MRI prostate — MRI and laboratory biomarkers
  Other Names: urine and blood biomarkers

SUMMARY:
The commercialization of MRI fusion biopsies has resulted in a dramatic increase in the use of MRI imaging for prostate cancer. How best to use MRI in the initial prostate biopsy setting given the availability of validated prostate cancer early detection markers is uncertain.This study will allow investigators to determine if prostate MRI is superior to validated panel of laboratory biomarkers (e.g. PCA3, PSA and TMPRSS2:ERG) in the initial biopsy setting.

DETAILED DESCRIPTION:
The primary aim of this study is to see if the addition of prostate MRI to a panel consisting of PSA, PCA3, TMPRSS2:ERG will significantly improve specificity for high-grade prostate cancer by 10%. The subsequent exploratory aims will 1) create an optimal panel of urine, blood and tissue biomarkers that will select those cases most likely to benefit from a MRI targeted biopsy, 2) directly compare PSA and urinary biomarkers with MRI to determine which ones are value added in the setting of initial biopsy, 3) evaluate changes in these biomarkers and MRI to determine if longitudinal changes predict subsequent high-grade prostate cancer, and 4) optimize MRI imaging to improve test performance. Importantly, this study will create a unique, prospective, cohort that will become the foundational reference set for of a range of future biomarker studies.

ELIGIBILITY:
Inclusion Criteria:

* Men with suspected but undiagnosed prostate cancer
* To be scheduled/scheduled for biopsy as routine clinical care

Exclusion Criteria:

* Inability to obtain blood and urine per SOP or conduct an attentive DRE
* Unable to undergo/tolerate a prostate MRI or failure to conduct the MRI
* Prior diagnosis of prostate cancer
* Prior prostate MRI unless being used as Index MRI (in this case index MRI can be one year prior to consent date)
* Participating in clinical trial for prostate disease
* Prior prostate surgery such as TURP, TUNA, TUMT, HOLEP, REZUM, UROlift
* Prior PCA3, TMPRSS2:erg or MIPS panel performed for clinical purpose

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology clinics
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinically significant prostate cancer | 2 years
  Pathologic diagnosis of prostate cancer with at least Gleason 7 or worse cancer grade on a needle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: John T Wei, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No